CLINICAL TRIAL: NCT04684459
Title: Phase I Study of Specific CAR-T Dual-targeting HER2 and PD-L1 for HER2-positive Solid Tumors
Brief Title: Dual-targeting HER2 and PD-L1 CAR-T for Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Director of Institute of Drug Clinical Trial of West China Hospital, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCART-002
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Peritoneal Carcinoma Metastatic; Pleural Effusion, Malignant; HER2 Positive Malignancies
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cell therapy (Experimental): Dual-targeting HER2 and PD-L1 CAR-T cell therapy
  Interventions: Biological: Dual-targeting HER2 and PD-L1 CAR-T cells

INTERVENTIONS:
Biological: Dual-targeting HER2 and PD-L1 CAR-T cells — HER2-positive solid tumor serosal cavity infusion

SUMMARY:
CAR-T therapy has achieved unprecedented success in hematological tumors in recent years, but the progress of CAR-T cells in the treatment of solid tumors is facing difficulties. HER-2 is frequently expressed in breast cancer, ovarian cancer, lung cancer, gastric cancer and other malignant tumors. In this study, the PD-L1 inhibitory signal was transformed into an activation signal in the tumor microenvironment, and enhanced the killing activity and survival ability of CAR-T cells. The HER-2/PD-L1 dual-targeting CAR-T will be investigated in patients with HER2-positive solid tumors, and all enrolled subjects will receive HER2/PD-L1 CAR T cells via intravenous or thoracic/peritoneal cavity infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, Age 18-75 years old; If the subjects are over 75 years old, the researchers will determine whether to enroll according to the basic health conditions of the subjects, regardless of gender. No upper age limit was set for chest/abdominal reinfusion CAR-T subjects.
2. Estimated life expectancy ≥ 3 months (according to investigator's judgement);
3. The Eastern Cooperative Oncology Group (ECOG) performance status score is 0-2;
4. Patients diagnosed as ovarian cancer, non-small cell lung cancer, breast cancer, gastric cancer, head and neck cancer, pancreatic cancer, colorectal cancer, transitional cell carcinoma, endometrial carcinoma, sarcoma, glioblastoma, cholangiocarcinoma, etc. have received standard systemic treatment, have systemic metastasis/serosal cavity metastasis or are not tolerated;
5. Expressing HER2 >20% of primary tumors or metastatic cells in the serous cavity by immunohistochemistry (IHC) or fluorescence in situ hybridization (FISH);
6. Absolute neutrophil count ≥ 1×10^9/L, platelet count ≥ 75×10^9/L, absolute lymphocyte count ≥0.5×10^8/L, hemoglobin ≥ 8.0 g/dl;
7. Creatinine clearance rate ≥60ml/min, Serum ALT/AST≤2.5 times of the normal level, and total bilirubin≤1.5 times of the normal level;
8. Cardiac ejection fraction ≥50%, no pericardial effusion;
9. No other serious diseases (autoimmune diseases or any immune deficiency disease or other disease in need of immunosuppressive therapy);
10. Patients must stop chemotherapy and targeted therapy for at least 3 weeks before starting treatment;
11. Patients must take reliable contraceptive measures before entering the trial, during the research process until 1 year after CAR-T infusion; reliable contraceptive measures will be determined by the main investigator or designated personnel;
12. Voluntarily participate in the research, understand and sign the informed consent;
13. The side effect of the last anti-tumor treatment was reduced to ≤1 grade, except for hair loss.

Exclusion Criteria:

1. Allergic to cytokines;
2. Uncontrolled activity infection;
3. Acute or chronic (graft-versus-host disease) GVHD;
4. Accompanied by other uncontrolled malignant tumors;
5. Patient with hepatitis B or C active period, HIV infection ≥ the upper limit of the normal level;
6. Suffer from serious diseases such as coronary heart disease, angina pectoris, myocardial infarction, arrhythmia, cerebral thrombosis, cerebral hemorrhage, etc.;
7. Patients with grade 2-3 hypertension or poorly controlled;
8. History of mental illness that is difficult to control;
9. Patients have used immunosuppressive agents for a long time after organ transplantation, except for recent or current inhaled corticosteroid therapy;
10. The existing medical history or mental state history or laboratory abnormalities may increase the risk associated with participating in the study or the administration of the study drug;
11. Unstable pulmonary embolism, deep venous embolism or other major arterial/venous thromboembolic events occurred within 6 months before enrollment. If receiving anticoagulant therapy;
12. Pregnant or nursing women, or plan to become pregnant during the treatment period or within 1 year after the treatment ends;
13. Patient suffering from diseases that have signed written informed consent or comply with research procedures; or are unwilling or unable to comply with research requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events | 12 months
  AE during the first 28 days after CAR-T cell administration
Dose-limiting toxicity (DLT) | 12 months
  Baseline up to 28 days after CAR-T cells infusion

SECONDARY OUTCOMES:
ORR（objective response rate） | Month 1，month 3, month 6
  Include CR（complete response）and PR（partial response）
DOR (duration of response) | 12 months
  The time from achievement of disease control

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Ma Q, He X, Zhang B, Guo F, Ou X, Yang Q, Shu P, Chen Y, Li K, Gao G, Zhu Y, Qin D, Tang J, Li X, Jing M, Zhao J, Mo Z, Liu N, Zeng Y, Zhou K, Feng M, Liao W, Lei W, Li Q, Li D, Wang Y. A PD-L1-targeting chimeric switch receptor enhances efficacy of CAR-T cell for pleural and peritoneal metastasis. Signal Transduct Target Ther. 2022 Nov 19;7(1):380. doi: 10.1038/s41392-022-01198-2. PMID 36402752